CLINICAL TRIAL: NCT01357460
Title: Endoscopic Lung Volume Reduction in Patients With Advanced Emphysema Due to alpha1 Antitrypsin Deficiency
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult patient recruitment
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Felix JF Herth, Prof. Dr. med. Felix Herth, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol D2.0 - 31.08.2010
Record Dates: First submitted 2011-05-16; First posted 2011-05-20 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hereditary Emphysema (Alpha 1-antitrypsin Deficiency)
Keywords: Emphysema; alpha1 antitrypsin deficiency; endoscopic lung volume reduction
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema

INTERVENTIONS:
Device: Implantation of intrabronchial valves (IBV) (Spiration IBV) — In advanced emphysema due to alpha1 antitrypsin deficiency even optimum treatment including drugs, physical training and possibly oxygen therapy is unable to influence exercise dyspnoea and exercise capacity.Implantation of intrabronchial valves in the most destroyed and hyperinflated lung lobe can improve the elastic recoil of the small airways by a reduction in lung volume and thus leading to more ergonomic breathing mechanics and diaphragm function.The one-way mechanism of these valves allows air to escape from the downstream lung segment without any influx of "new" air during inspiration.
  Other Names: Spiration IBV

SUMMARY:
Patients with advanced heterogeneous emphysema due to alpha1 antitrypsin deficiency might benefit from endoscopic implantation of intrabronchial valves.

DETAILED DESCRIPTION:
Patient enrollment and data acquisition is to be carried out on a prospective basis. It is planned to enroll a total of 25 patients with advanced heterogeneous emphysema due to alpha1 antitrypsin deficiency. All patients will undergo treatment at one study centre in Heidelberg. Therapy of all patients consists of implantation of intrabronchial valves (IBV, Spiration, Olympus) in the most emphysematous destroyed lobe.

ELIGIBILITY:
Inclusion Criteria:

* pulmonary function: FEV1 < 45 %, RV > 150 %, TLC > 100 %
* alpha1 antitrypsin deficiency (< 80 mg/dl), genotype: PiZS, PiZZ, Pi0/0
* heterogenous emphysema

Exclusion Criteria:

* homogenous emphysema
* significant bronchiectasis
* severe concomitant diseases
* pregnancy

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-09-24 (Actual); Study Completion 2014-12-30 (Actual)

PRIMARY OUTCOMES:
Improvement in pulmonary function (FEV1 (forced expiratory volume in 1 second) and RV/TLC (residual volume/total lung capacity) | 3 months

SECONDARY OUTCOMES:
Number of major complications | 3 months
Evaluation of IBV migration rate | 3 months
Average changes in pulmonary function (FEV1, VC (vital capacity), RV, TLC, RV/TLC) | 3 months
Average changes in 6-minute-walk-distance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Gompelmann, MD, Principal Investigator — Heidelberg University
Locations (1):
- Thoraxklinik, Heidelberg, Germany